CLINICAL TRIAL: NCT04253808
Title: Feasibility of a Carbohydrate-restricted, High-fat Diet to Improve Outcomes in Head and Neck Squamous Cell Carcinoma: A Pilot Randomized Controlled Feeding Trial
Brief Title: Feasibility of a Carbohydrate-restricted, High-fat Diet on Head and Neck Squamous Cell Carcinoma Outcomes
Acronym: CRHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Augusta Victoria Hospital, East Jerusalem (Unknown)
Responsible Party: Principal Investigator, Anna Arthur, Assistant Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19635
Record Dates: First submitted 2020-01-15; First posted 2020-02-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: non-metastatic
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Diet, High-Fat

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: Participants will be blinded from the group they are assigned to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): The experimental arm (N=6) were provided a CRHF diet with enough calories to maintain body weight for appoximately 2 weeks neoadjuvantly (during radiotherapy preparation) and adjuvantly during primary oncology treatment for ~6.5 weeks. The CRHF diet was composed of 45% fats (mostly) unsaturated fats, 25% proteins, and 30% carbohydrates.
  Interventions: Behavioral: Carbohydrate-restricted, high-fat diet
- Arm B (Active Comparator): Arm B (N=7) were provided a regular composition diet prescribed with enough calories to maintain body weight for approximately 2 weeks neoadjuvantly (during radiotherapy preparation) and adjuvantly during primary oncology treatment for ~6.5 weeks.
  The regular composition diet was composed of ~50-52% carbohydrates, ~30% fats, and 18-20% proteins,
  Interventions: Behavioral: Regular composition diet
- Control group (No Intervention): The control group (N=26) followed applicable eligibility criteria but did not receive any intervention.

INTERVENTIONS:
Behavioral: Carbohydrate-restricted, high-fat diet — Diet composition was ~45% fats, ~30% carbohydrates, and ~25% proteins. Calorie needs were provided according to what the Bioelectrical Impedance (BIA) device gave as required to maintain bodyweight.
  Sources of macronutrients:
  * Carbohydrates: from whole grains, dairy products, legumes, fruits, and vegetables.
  * Fats: from mono- and polyunsaturated fatty acids, including medium- and long-chain fatty acids.
  * Proteins: plant-based proteins and lean animal-based proteins. All meals were provided to the participants throughout the study period and the diet was provided orally unless the patient was on a feeding tube or a feeding tube is ordered by a physician during the study period. Diet texture was according to patients chewing and swallowing abilities. If the patient is on a feeding tube or intake is insufficient, a formula with similar macronutrient composition + a protein supplement was provided.
  Other Names: CRHF diet
  Arms: Arm A
Behavioral: Regular composition diet — The regular composition diet contained approximately 50-52% carbohydrates, 30% fats, and 18-20% proteins
  Arms: Arm B

SUMMARY:
This study will test the feasibility of a carbohydrate-restricted, high-fat (CRHF) diet intervention in newly diagnosed head and neck squamous cell carcinoma patients who will receive definitive radiation.

DETAILED DESCRIPTION:
Our previous observational research indicates that a pretreatment diet high in total carbohydrates is associated with increased risk of all-cause and disease-specific mortality in head and neck cancer. The purpose of this study is to conduct a single-blinded randomized controlled trial to test the feasibility of a carbohydrate-restricted, high-fat (CRHF) diet intervention in newly diagnosed head and neck cell squamous carcinoma (HNSCC) patients who will receive definitive radiation. The secondary aim is to collect preliminary data on the effect of the intervention on tumor progression, nutritional status, body composition, quality of life, and symptom burden.

Thirteen newly diagnosed HNSCC non-metastatic patients were recruited from Augusta Victoria Hospital in East Jerusalem and randomized into one of two arms; a carbohydrate-restricted, high-fat diet arm (arm A) and a regular diet composition arm (Arm B). Arm A (N=6) were provided a CRHF diet both neoadjuvantly (for 2 weeks prior to treatment) and adjuvantly (during treatment with radiation). Arm B (N=7) received standard oncologic treatment including a regular diet (50-52% carbohydrates, 30% fats, and 18-20% proteins). Feasibility outcomes, including recruitment, retention, intervention adherence, and safety were tracked weekly. Biomarkers, tumor progression, nutritional status, body composition, QOL, and symptoms were assessed at baseline, 2-weeks, and 2-3 months post-treatment. A control group (N=26) included HNSCC patients who follow the same applicable eligibility criteria and did not receive any kind of dietary intervention. Medical information were collected retrospectively from the control group patients' files. Information on demographics (age, sex, smoking status, weight, height, marital status, education, occupation, and residency), tumor site, cancer stage, treatment dose reduction, treatment break, early cessation of treatment, hospitalization, symptoms, and weight loss, were collected during treatment from arms A and B and retrospectively from the control group.

This proposed pilot/feasibility study is the first step in determining if a CRHF diet is an effective treatment modality in cancer and if providing a diet with any composition before and during treatment is more beneficial than not providing a diet at all.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed with non-metastatic cancer of the oral cavity, hypopharynx, oropharynx, or larynx
2. Plan to receive definitive radiation treatment at Augusta Victoria Hospital (AVH) in East Jerusalem
3. Age > 18
4. Karnofsky Index of ≥70 %
5. Normal liver and kidney function tests
6. Able to understand and willingly sign a written informed consent document
7. Lives in the West Bank or Gaza
8. Has an oven/microwave and a refrigerator where they are staying
9. Cancer stage 1-4 with no metastasis
10. BMI > 20 kg/m²

Exclusion Criteria:

1. Those who do not meet the inclusion criteria
2. Have metastatic disease
3. Will receive a palliative treatment
4. On insulin treatment or other diabetic treatment
5. Uncontrolled illness (e.g. active infection, symptomatic CHF, cardiac arrhythmia, or psychiatric illness)
6. Received previous treatment for another primary cancer
7. Diagnosed with an illness that requires dietary modifications (e.g. renal disease, liver disease, celiac disease, and inflammatory bowel disease)
8. Already consuming a carbohydrate-restricted, high-fat diet
9. On chronic system corticosteroids for any reason (inhaled corticosteroids are allowed);
10. Pregnant or lactating women
11. Body mass index (BMI) < 20
12. Will start treatment within <2 weeks from screening day
13. Requires parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Feasibility measure: Recruitment | Through study completion, an average of 2 years
  Recruitment will be measured by recording the number of patients screened, included, excluded, dropped-out, and completed the study throughout the study period.
Feasibility measure: Adherence | Throughout the 16.5 week study period (from baseline till the end of study)
  Adherence will be measured by collecting daily food surveys that ask about daily food intake (checking the food items that have been consumed and providing information about any other additional foods that were consumed) as well as completing all study activities which are listed on a checklist.
Feasibility measure: Retention | Throughout 16.5 week study period (from baseline till the end of study)
  Retention will be measured by recording the number of patients included or agreed to participate and completed all study protocol.
Blood Glucose | Throughout the 8.5 weeks of intervention
  Blood glucose level was measured, recorded, and mentioned whether the level was normal, low, or high.
Complete blood count (CBC) | Throughout the 8.5 weeks of intervention
  CBC levels were measured, recorded, and mentioned whether levels were normal, low, or high.
Liver function | Throughout the 8.5 weeks of intervention
  Liver function tests were measured, recorded, and mentioned whether levels were normal, low, or high. These tests were done to assess whether liver function remained normal after consuming the diet or not. That was done by measuring the levels of GOT, GPT, and alkaline phosphatase in the blood and recording whether they were normal or not.
Kidney function | Throughout the 8.5 weeks of intervention
  Kidney function tests were measured, recorded, and mentioned whether levels were normal, low, or high. These tests were done to assess whether kidney function remained normal after consuming the diet or not. That was done by measuring the levels of BUN, creatinine, and uric acid in the blood and recording whether they were normal or not.
Potassium | Throughout the 8.5 weeks of intervention
  Potassium level was measured, recorded, and mentioned whether the level was normal, low, or high.
Phosphorus level was measured, recorded, and mentioned whether the level was normal, low, or high. | Throughout the 8.5 weeks of intervention
  Phosphorus
Magnesium | Throughout the 8.5 weeks of intervention
  Magnesium level was measured, recorded, and mentioned whether the level was normal, low, or high.
Sodium | Throughout the 8.5 weeks of intervention
  Sodium level was measured, recorded, and mentioned whether the level was normal, low, or high.
Chloride | Throughout the 8.5 weeks of intervention
  Chloride level was measured, recorded, and mentioned whether the level was normal, low, or high.
Calcium | Throughout the 8.5 weeks of intervention
  Calcium level was measured, recorded, and mentioned whether the level was normal, low, or high.
Albumin level | Throughout the 8.5 weeks of intervention
  Albumin level was measured, recorded, and mentioned whether the level was normal, low, or high.
C-reactive protein (CRP) level | Throughout the 8.5 weeks of intervention
  CRP level was measured, recorded, and mentioned whether the level was normal, low, or high. High level indicates inflammation.
Total protein level | Throughout the 8.5 weeks of intervention
  Total protein level was measured, recorded, and mentioned whether the level was normal, low, or high.
Insulin level | Throughout the 8.5 weeks of intervention
  Insulin level was measured, recorded, and mentioned whether the level was normal, low, or high.
Triglycerides level | Throughout the 8.5 weeks of intervention
  Triglycerides levels were measured, recorded, and mentioned whether the levels were normal, low, or high.
Total cholesterol level | Throughout the 8.5 weeks of intervention
  Total cholesterol level was measured, recorded, and mentioned whether the level was normal, low, or high.
LDL-cholesterol level | Throughout the 8.5 weeks of intervention
  LDL-cholesterol level was measured, recorded, and mentioned whether the level was normal, low, or high.
HDL-cholesterol level | Throughout the 8.5 weeks of intervention
  HDL-cholesterol level was measured, recorded, and mentioned whether the level was normal, low, or high.

SECONDARY OUTCOMES:
Tumor progression assessment | Throughout 16.5 week study period (from baseline till the end of study)
  Tumor progression was assessed using RECIST and WHO criteria as well as diagnostic CTScan/ PETScan imaging.
Nutritional status assessment | Throughout 16.5 week study period (from baseline till the end of study)
  Nutritional status was assessed using the "Patient generated subjective global assessment" (PG-SGA) tool.
Percentage of body fat | Throughout 16.5 week study period (from baseline till the end of study)
  The percentage of body fat was measured by using a Bioelectric Impedance Analysis (BIA) device and used to study the effect of the intervention on body composition.
Percentage of lean body mass | Throughout 16.5 week study period (from baseline till the end of study)
  The percentage of lean body mass was measured by using a Bioelectric Impedance Analysis (BIA) device and used to study the effect of the intervention on body composition.
Percentage of body water | Throughout 16.5 week study period (from baseline till the end of study)
  The percentage of body water was measured by using a Bioelectric Impedance Analysis (BIA) device and used to study the effect of the intervention on body composition.
Basal metabolic rate (BMR) | Throughout 16.5 week study period (from baseline till the end of study)
  BMR was measured by using a Bioelectric Impedance Analysis (BIA) device and used to study the effect of the intervention on body composition.
Quality of life assessment | Throughout 16.5 week study period (from baseline till the end of study)
  Quality of life was assessed using EORTC QLQ questionnaires.
Symptom burden assessment | Throughout 16.5 week study period (from baseline till the end of study)
  Symptom burden was assessed using the validated Memorial Symptom Assessment Survey.
Hospitalization | Throughout the 8.5 weeks of intervention
  We recorded whether the participant was hospitalized or not.
Number of hospitalizations | Throughout the 8.5 weeks of intervention
  If the participant was hospitalized, we recorded the number of hospitalizations
Duration of hospitalization | Throughout the 8.5 weeks of intervention
  If the participant was hospitalized, we recorded the duration of each hospitalization
Weight loss | Throughout 16.5 week study period (from baseline till the end of study)
  We recorded whether the participant had weight loss or not
Amount and span of weight loss | Throughout 16.5 week study period (from baseline till the end of study)
  If the participant had weight loss, we recorded how much he had lost and during what time span
Treatment dose reduction | Throughout the 6.5 weeks of treatment
  We recorded whether there was treatment dose reduction and the reason for that.
Treatment break | Throughout the 6.5 weeks of treatment
  We recorded whether there was treatment break and the reason for that.
Early cessation of treatment | Throughout the 8.5 weeks of treatment
  We recorded whether there was early cessation of treatment and the reason for that.

CONTACTS AND LOCATIONS:
Overall Officials: Anna E Arthur, PhD, MPH, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Augusta Victoria Hospital, East Jerusalem, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No
To learn more about this study, you or your doctor may contact the study research staff using the contact information provided by the sponsor.

REFERENCES:
- [Background] Arthur AE, Goss AM, Demark-Wahnefried W, Mondul AM, Fontaine KR, Chen YT, Carroll WR, Spencer SA, Rogers LQ, Rozek LS, Wolf GT, Gower BA; University of Michigan Head and Neck SPORE Program. Higher carbohydrate intake is associated with increased risk of all-cause and disease-specific mortality in head and neck cancer patients: results from a prospective cohort study. Int J Cancer. 2018 Sep 1;143(5):1105-1113. doi: 10.1002/ijc.31413. Epub 2018 Apr 17. PMID 29604042